CLINICAL TRIAL: NCT04200625
Title: Effects of Semaglutide vs Dulaglutide on Epicardial Adipose Tissue Thickness in Subjects With Type 2 Diabetes and Obesity
Brief Title: Semaglutide vs Dulaglutide on Epicardial Adipose Tissue
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Medicine, University of Miami
Other Study IDs: 20190944
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Epicardial Fat

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Semaglutide: Patients using standard of care weekly GLP-1A analog Semaglutide
- Dulaglutide: Patients using standard of care weekly GLP-1A analog Dulaglutide
- Metformin: Patients using standard of care daily Metformin.

SUMMARY:
Epicardial Fat (EAT), the visceral fat depot of the heart, is a modifiable cardio-metabolic risk factor and therapeutic target. EAT expresses GLP-1 receptors (GLP-1R). GLP-1 receptor agonist liraglutide is known to significantly decrease EAT thickness. However, the effects of GLP-1 receptor agonists semaglutide and dulaglutide on EAT thickness are unknown

DETAILED DESCRIPTION:
This is a retrospective, observational, case control study. Data were obtained from retrospective review of the electronic medical records.

Patients were treated with either semaglutide, dulaglutide or metformin as standard of care, during routine clinical practice, regardless of the study. Each patient underwent routine labs and an onsite ultrasound measurement of EAT thickness at baseline and at the routine 12-week follow up visit, as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes,
* BMI ≥27 kg/m2,
* Age ≥ 18 years old

Exclusion Criteria:

* Type 1 diabetes
* Concurrent use of dipeptidyl peptidase 4 (DPP-4) inhibitors or other GLP-1 agonist receptors
* History of diabetic ketoacidosis
* Known contraindications to GLP-1 receptor agonists such as previous history of pancreatitis or medullary thyroid carcinoma, personal or family history of multiple endocrine neoplasia type 2
* Acute infective diseases, cancer or chemotherapy
* Use of systemic corticosteroids within the 3 months prior this study
* Known or suspected allergy to semaglutide or dulaglutide excipients or related products
* Pregnancy, breastfeeding or the intention of becoming pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic subjects who routinely come to the University of Miami Division of Diabetes, Endocrinology and Metabolism outpatient diabetic clinic, as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Epicardial Fat thickness | 12 weeks
  Ultrasound measured Epicardial Fat thickness

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Iacobellis, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No